CLINICAL TRIAL: NCT00730106
Title: Endoscopic Findings in Taiwan Patients Presenting With Characteristic Symptoms of Gastroesophageal Reflux Disease
Brief Title: Endoscopic Findings in Patients With Typical Gastroesophageal Reflux Disease (GERD) Symptoms
Status: Completed | Type: Observational
Sponsor: Lotung Poh-Ai Hospital (Other)
Responsible Party: Hsing-Hong Chen/Superintendent, Lotung Poh-Ai hospital
Other Study IDs: OMCP-97-017
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal reflux disease; Alarm symptoms; Gastrointestinal endoscopy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Patients with pre-defined alarm symptoms
- 2: Patients without pre-defined alarm symptoms

SUMMARY:
Gastroesophageal reflux disease (GERD) is diagnosed on the basis of characteristic reflux symptoms (i.e. troublesome heartburn and/or acid regurgitation). Empirical therapy without diagnostic endoscopy is suggested for those GERD patients presenting without alarm symptoms in Western countries. Whether such "treating instead of testing" strategy should be applied in Asia, an area with higher prevalence of Helicobacter pylori and gastric cancer, remains uninvestigated.

DETAILED DESCRIPTION:
This study amis to investigate upper endoscopic findings of typical acid reflux patients with and without alarm symptoms in Taiwan During the period from May 2008 to December 2009, consecutive adult outpatients, who receive upper endoscopy for characteristic reflux symptoms of heartburn or acid regurgitation, are invited to participate. All study participants are evaluated for presence of pre-defined alarm symptoms including odynophagia or dysphagia, gastrointestinal bleeding, involuntary body weight loss and anemia.

Upper endoscopic procedures are performed with standard electronic videoendoscope (GIF-Q240 or GIF-Q260; Olympus, Tokyo, Japan) by experienced endoscopists; each of them had previously performed a minimum of 2,000 upper endoscopy exams. Representative images are taken and stored as electronic files in a digital image system for later analysis.

The following five significant endoscopic findings are pre-defined endpoints of this study: 1) any malignant lesion in the upper digestive tract, 2) Barrett esophagus, 3) severe erosive esophagitis (LA grade C or D), 4) peptic stricture, 5) peptic ulcer.

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* chief complaints of characteristic GERD symptoms (heart burn or acid regurgitation), evaluated by standard questionnaire
* undergo upper digestive endoscopy

Exclusion Criteria:

* age less than 18 years old or more than 90 years old
* unable to complete upper endoscopy
* known diagnosis of gastroesophageal malignancy
* follow-up visit for known gastroesophageal lesion identified by previous upper endoscopy
* failure to obtain informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult outpatients with characteristic GERD symptoms, in a district general hospital
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pre-defined significant upper digestive endoscopic findings | within one month after the endoscopy examination

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Chun Hsu, M.D., Principal Investigator — Lotung Poh-Ai Hospital
Locations (1):
- Lotung Poh-Ai Hospital, Lotung Town, Ilan County, Taiwan